CLINICAL TRIAL: NCT02353598
Title: A Phase Ib, Multicenter, Randomized, Placebo-Controlled, Double-Blind, Parallel-Arm, Multiple-Dose Study to Assess The Safety, Tolerability, And Pharmacokinetics of Intravenous Crenezumab Administered in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: A Study of Crenezumab in Participants With Mild to Moderate Alzheimer Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GN29632
Record Dates: First submitted 2015-01-23; First posted 2015-02-03 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Double-blind treatment window: Crenezumab dose level 1 (Experimental): Participants will recieve crenezumab dose level 1 once every 4 weeks.
  Interventions: Drug: Crenezumab dose level 1
- Double-blind treatment window: Crenezumab dose level 2 (Experimental): Participants will receive crenezumab dose level 2 once every 4 weeks.
  Interventions: Drug: Crenezumab dose level 2
- Double-blind treatment window: Crenezumab dose level 3 (Experimental): Participants will receive crenezumab dose level 3 once every 4 weeks.
  Interventions: Drug: Crenezumb dose level 3
- Double-blind treatment window: Placebo (Placebo Comparator): Participants will receive placebo matched to crenezumab once every 4 weeks.
  Interventions: Drug: Placebo
- Optional OLE window: Crenezumab (Experimental): Participants will receive crenezumab dose levels 1 2, or 3 once in every 4 weeks.
  Interventions: Drug: Crenezumab dose level 1; Drug: Crenezumab dose level 2; Drug: Crenezumb dose level 3

INTERVENTIONS:
Drug: Crenezumab dose level 1 — Participants will receive crenezumb dose level 1 IV infusion once every 4 weeks up to Week 13 in double-blind treatment window or up to Week 61 in optional OLE window.
  Arms: Double-blind treatment window: Crenezumab dose level 1; Optional OLE window: Crenezumab
Drug: Crenezumab dose level 2 — Participants will receive crenezumb dose level 2 IV infusion once every 4 weeks up to Week 13 in double-blind treatment window or up to Week 61 in optional OLE window.
  Arms: Double-blind treatment window: Crenezumab dose level 2; Optional OLE window: Crenezumab
Drug: Crenezumb dose level 3 — Participants will receive crenezumb dose level 3 IV infusion once every 4 weeks upto Week 13 in double-blind treatment window or up to Week 61 in optional OLE window.
  Arms: Double-blind treatment window: Crenezumab dose level 3; Optional OLE window: Crenezumab
Drug: Placebo — Participants will receive placebo matched to crenezumab IV infusion once every 4 weeks upto Week 13 in double-blind treatment window.
  Arms: Double-blind treatment window: Placebo

SUMMARY:
This randomized, placebo-controlled, double-blind, parallel-arm study will evaluate the safety and tolerability of at least two dose levels of intravenous (IV) crenezumab in 24-72 participants with mild to moderate Alzheimer disease (AD) (mini-mental state examination [MMSE] 18 to 28 points, inclusive). An optional open-label extension (OLE) will be offered after the completion of initial double-blind stage.

ELIGIBILITY:
Inclusion Criteria:

* Body weight greater than or equal (>/=) 45 kilograms (kg) and less than or equal (</=) 120 kg
* Ages 50-90 years, inclusive
* Availability of a person ("caregiver") who, in the investigator's judgment, has frequent and sufficient contact with the participant and is able to provide accurate information regarding the participant's cognitive and functional abilities, agrees to provide information at clinic visits, which require partner input for scale completion, and signs the necessary consent form
* Willingness and ability to complete all aspects of the study; the participant should be capable of completing assessments either alone or with the help of the caregiver
* Adequate visual and auditory acuity, in the investigator's judgment, sufficient to perform the neuropsychological testing
* Clinical diagnosis of probable mild to moderate AD based on the national institute on neurological and communication disease and stroke/Alzheimer's disease and related disorders association (NINCDS/ADRDA) criteria or probable major neurocognitive disorder due to AD of mild to moderate severity based on diagnostic and statistical manual of mental disorders, version 5 (DSM-5) criteria
* Screening MMSE score of 18-28 points, inclusive
* Screening clinical dementia rating global score (CDR-GS) of 0.5 or 1.0
* Screening geriatric depression (GDS)-15 score less than (<) 6
* Positive florbetapir amyloid positron emission tomography (PET) scan by qualitative read conducted by the core/central PET laboratory
* Women must be postmenopausal or surgically sterile
* Men with female partners of childbearing potential agree to remain abstinent or use adequate methods of contraception as defined by protocol during the treatment period and for at least 8 weeks after the last dose of study drug and agreement to refrain from donating sperm during this same period

Exclusion Criteria:

* History or presence of clinically evident vascular disease potentially affecting the brain that, in the opinion of the investigator, has the potential to affect cognitive function
* History or presence of stroke within the previous 2 years or documented history of transient ischemic attack within the previous 12 months
* History of severe, clinically significant central nervous system trauma
* History or presence of intracranial tumor that is clinically relevant in the opinion of the investigator
* Presence of infections that affect brain function or history of infections that resulted in neurologic sequelae
* History or presence of systemic autoimmune disorders potentially causing progressive neurologic disease with associated cognitive deficits
* History or presence of a neurologic disease other than AD that may affect cognition
* Presence of superficial siderosis, more than four cerebral microhemorrhages, or evidence of a prior cerebral macrohemorrhage
* Inability to tolerate magnetic resonance imaging (MRI) procedures or contraindication to MRI
* History or presence of atrial fibrillation except if only one episode that resolved more than 1 year ago and for which treatment is no longer indicated or that in the investigator's judgment poses no risk for future stroke
* Within the previous 2 years, unstable or clinically significant cardiovascular disease
* Uncontrolled hypertension
* Chronic kidney disease of Stage >/= 4, according to the national kidney foundation kidney disease outcomes quality initiative (NKF KDOQI) guidelines for chronic kidney disease
* Impaired hepatic function
* Clinically significantly abnormal screening blood or urine that remain abnormal on retest
* History of malignancies within 5 years prior to screening, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer; cancer that is considered likely to be cured, is not being actively treated with anti-cancer therapy or radiotherapy and not likely to require treatment in the ensuing 5 years as well as cancers that are considered to have low probability of recurrence are allowed
* Known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human, or humanized antibodies or fusion proteins
* Severe or unstable medical condition that, in the opinion of the investigator or sponsor, could be expected to progress, recur, or change to such an extent that it could put the patient at special risk, bias the assessment of the clinical or mental status of the patient to a significant degree, interfere with the patient's ability to complete the study assessments, or would require the equivalent of institutional or hospital care
* Any previous treatment with medications used to treat Parkinsonian symptoms or any other neurodegenerative disorder within 1 year before screening even if the patient is taking the medicine for a non-neurodegenerative disorder such as restless leg disorder
* Typical anti-psychotic or neuroleptic medication within 6 months before screening except as brief treatment for a non-psychiatric indication
* Antihemostasis medication within 2 weeks before screening
* Sedative, hypnotic, or benzodiazepine medication within 3 months before screening except intermittent use of the following for sleep or anxiety: alprazolam, lorazepam, oxazepam, temazepam, diazepam, or a short-acting benzodiazepine-like medication

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-02-26 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Number of participants with anti-crenezumab antibodies | From baseline up to follow-up period (Week 69)
Number of participants with suicidal ideation, suicidal behavior, and self-injurious behavior without suicidal intent, as determined using the columbia-cuicide severity rating scale (C-SSRS) | From baseline up to follow-up period (Week 69)
Number of participants with changes from baseline in vital signs, electrocardiogram (ECG) and clinical laboratory results | From baseline up to follow-up period (Week 69)
Number of participants with amyloid-related imaging abnormalities-hemorrhage (ARIA-H) | Up to Week 13
Number of participants with adverse events (AEs) and serious adverse events (SAEs) according to national cancer institute common terminology criteria for adverse events, version 4.0 (NCICTCAE v4.0) | From baseline up to follow-up period (Week 69)
Number of participants with of non-serious AEs of special interest | From baseline up to follow-up period (Week 69)
Number of participants with amyloid-related imaging abnormalities-edema/effusion (ARIA-E) | Up to Week 13

SECONDARY OUTCOMES:
Serum concentration of crenezumab | Pre-dose on Day 1, 60-90 minutes (min) post infusion on Day 1, Days 2, 8, Week 2, pre-dose and 60-90 min post infusion on dosing day of Weeks 5, 9, 13, and 21; pre-dose and 60-90 min post infusion on dosing day of Weeks 25, 53, 61, and 69

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- United States (13):
  - Mayo Clinic Scottsdale, Phoenix, Arizona
  - UCSF - Memory and Aging Center, San Francisco, California
  - Brain Matters Research, Inc., Delray Beach, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Bioclinica Orlando, Orlando, Florida
  - Bioclinica The Villages, The Villages, Florida
  - Indiana University School Of Medicine; Department Of Neurology, Indianapolis, Indiana
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Millennium Psychiatric Associates, LLC, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - UNiversity of Rochester, Rochester, New York
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Roper St. Francis Healthcare; Clinical Biotechnology Research Institute, Charleston, South Carolina

REFERENCES:
- [Derived] Guthrie H, Honig LS, Lin H, Sink KM, Blondeau K, Quartino A, Dolton M, Carrasco-Triguero M, Lian Q, Bittner T, Clayton D, Smith J, Ostrowitzki S. Safety, Tolerability, and Pharmacokinetics of Crenezumab in Patients with Mild-to-Moderate Alzheimer's Disease Treated with Escalating Doses for up to 133 Weeks. J Alzheimers Dis. 2020;76(3):967-979. doi: 10.3233/JAD-200134. PMID 32568196
- [Derived] Yoshida K, Moein A, Bittner T, Ostrowitzki S, Lin H, Honigberg L, Jin JY, Quartino A. Pharmacokinetics and pharmacodynamic effect of crenezumab on plasma and cerebrospinal fluid beta-amyloid in patients with mild-to-moderate Alzheimer's disease. Alzheimers Res Ther. 2020 Jan 22;12(1):16. doi: 10.1186/s13195-020-0580-2. PMID 31969177